CLINICAL TRIAL: NCT03875625
Title: Change of Adipose Tissues and Triglyceride in Obese Patients With Non-alcoholic Fatty Liver Disease After Bariatric Surgery or Life-style Intervention
Brief Title: Change of Adipose Tissues and Triglyceride After Bariatric Surgery or Life-style Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Winnie W.C. Chu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018.612
Record Dates: First submitted 2019-03-08; First posted 2019-03-15 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Obesity, Morbid; Brown Fat; Metabolic Disease; Diabetes Mellitus; Insulin Resistance; Abdominal Subcutaneous Fat
Keywords: MRI; Dietitian Lifestyle intervention; Bariatric surgery; Brown adipose tissue; White adipose tissue; no alcoholic fatty liver disease; diabetes mellitus type 2; Pancreatic fat
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity, Morbid; Metabolic Diseases; Diabetes Mellitus; Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Four groups of interventional groups will be applied. Group 1 for subjects with morbid obesity who have consented to bariatric surgery, Group 2 for subjects with morbid obesity and have opted for dietitian led lifestyle modification intervention, Group 3 and 4 for subjects with mild to moderate obesity randomly (RCT) assigned to either dietitian led life style modification intervention group or conventional care (control group).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Morbid obesity- Bariatric surgery group (Experimental): Morbid obese subjects who will consent to bariatric surgery
  Interventions: Procedure: Bariatric surgery
- Morbid obesity-Dietitian led life style intervention group (Experimental): Morbid obese subjects who will not consent to bariatric surgery but instead opt for dietitian led life style intervention
  Interventions: Behavioral: Dietitian led life style modification intervention
- Mild obesity-Dietitian led life style intervention group (Experimental): Mild- Moderate subjects assigned through a randomized controlled trial to the dietitian led life style intervention
  Interventions: Behavioral: Dietitian led life style modification intervention
- Mild obesity-Conventional care group (control) (Experimental): Mild- Moderate subjects assigned through a randomized controlled trial to conventional care
  Interventions: Behavioral: Conventional care (control)

INTERVENTIONS:
Procedure: Bariatric surgery — Use of the normal bariatric surgery procedures commonly conducted in our hospital, such as: Laparoscopic Roux-en-Y gastric bypass (RYGB) and Laparoscopic sleeve gastrectomy (LSG)
  Arms: Morbid obesity- Bariatric surgery group
Behavioral: Dietitian led life style modification intervention — Intensive 6 months life style changes supervised by diatitians.
  Arms: Mild obesity-Dietitian led life style intervention group; Morbid obesity-Dietitian led life style intervention group
Behavioral: Conventional care (control) — receive routine care
  Arms: Mild obesity-Conventional care group (control)

SUMMARY:
The study is aimed

* To quantify the change of adipose tissues, triglyceride in liver and pancreas and cholesterol after lifestyle intervention or bariatric surgery.
* To test the hypothesis that Brown fat is an independent biomarker for the development of Non Alcoholic Fat Liver Disease (NAFLD)
* To study the association among Brown fat, NAFLD and obesity.

DETAILED DESCRIPTION:
Obesity is associated with different chronic disorders such as metabolic syndrome, non-alcoholic fatty liver disease (NAFLD) and diabetes mellitus type 2 (DM2). It can be classified into mild, moderate and severe using different cut-off values of body mass index (BMI). Many interventions and treatments against obesity have been proposed. Patients with mild to moderate obesity are suggested to undergo lifestyle monitoring or intervention programs while patients with severe or morbid obesity may be suggested to undergo bariatric surgery. Brown adipose tissue (BAT) is a specific type of adipose tissue with unique ability to produce heat by non-shivering thermogenesis. It increases energy expenditure and lower blood glucose levels and therefore it is suggested to be a potential therapy against obesity, NAFLD, DM2 etc.

Research studies demonstrated that obesity is strongly associated with NAFLD. From our previous observation, most obese individuals suffer from NAFLD. Nevertheless, a small portion of them are protected from NAFLD. We try to understand why and how this small portion of severe obese patients can keep themselves protected from NAFLD while some lean individual suffers from it. We would also like to test whether the amount of BAT is a biomarker for NAFLD. Besides, we would like to validate the accuracy of liver inflammation and fibrosis (LIF) scores with liver biopsy results.

The change of adipose tissues (i.e. brown, subcutaneous, visceral), triglyceride in liver and pancreas and cholesterol (i.e. HDL and LDL) in bloodstream would be measured in patients with NAFLD who undergo either bariatric surgery or lifestyle intervention. 40 subjects will be recruited. Half of them for the lifestyle intervention group while half for the bariatric group. Baseline MRI and blood test will be performed before the start of their treatments and two follow-up scans as well as blood tests in six-month and twelve-month intervals.

This study allows objective measurement to evaluate efficacy of different treatments against obesity and the response of NAFLD after weight loss. Furthermore, this study provides quantitative measurement of BAT and tests whether BAT is associated with NAFLD or other metabolites disorders such as DM2 and hyperlipidemia.

b) Research plan and methodology Subjects Eighty volunteers will be recruited for this project. 40 of them with mild-moderate obesity and the other 40 subjects with morbid obesity.

Morbid obesity subjects will be further divided into bariatric group (those who gave consent for surgery i.e. 20 subjects and 20 for lifestyle intervention group.

The mild- moderate obesity group will also be divided into two subgroups (20 in each group) through a randomization process in a 1:1 ratio to participate in the dietitian led life style modification program or receive usual care. The computer will be used to generate a list of random numbers for randomization of the two groups and this will be done in blocks of six by Nursing officers working in the clinic. The treatment assignments will be concealed in numbered sealed envelopes which will only be opened sequentially upon patient enrollment. Blinding methods to treatment assignments will be employed to both clinicians and radiographers during analysis and patient assessments. Inclusion criteria involve individuals between the age of 18-65, BMI ≥ 25-30 kg/m2 for mild-moderate obesity, BMI ≥ 30 kg/m2 with metabolic syndrome or BMI ≥ 35 kg/m2 for morbid obesity, who have been diagnosed with NAFLD. Exclusion criteria include other kind of hepatic diseases or under medications that are known to affect liver fat accumulation, weight≥250 kg, waist circumference≥150 cm. The maximum weight and waist circumference are set due to the tolerance of the scanner and its bore size. Written informed consents will be obtained from all volunteers.

Protocol The protocol in this part of the study will be as described by Wong et al. At the commencement of the study, all the 80 patients will initially be assessed by the dietitian and relevant individual recommendations will be provided. This will include complete behavioral change assessments, covering important areas such as the patient's current eating habits, lifestyles patterns etc.

Surgical group (bariatric surgery) The surgical group will be identified from the surgical team and will be enrolled by the surgical team accordingly.

Lifestyle Modification Group Patients randomized to the intervention group will participate in a dietitian-led lifestyle modification programme for 12 months. The programme will be held at 2 urban centres that are open to the public for the management of obesity and related disorders. The programme will be based on a strategy of increasing energy expenditure and reducing caloric intake using lifestyle behavioral change to achieve long-lasting impact. The patients will attend dietary consultation sessions weekly in the first 4 months, and monthly in the following 8 months. At the first session (about 1 h), the dietitian will carry out a complete behavioral assessment, covering important areas such as the patient's current eating and lifestyle patterns, specific eating-related behaviors, knowledge of risks associated with current eating patterns, concerns and feelings about specific lifestyle changes. The dietitian will also discuss the expected duration and specific dietary and lifestyle advices to achieve a desirable weight status with the patients.

In the follow-up sessions (about 20 minutes), the dietitian will review the patient's dietary practice and provide recommendations. Each patient will be given an individualized menu plan. The dietary component and portion sizes of the menu plan will be based on the recommendations of the American Dietetic Association . A varied balanced diet with an emphasis on fruit and vegetables, and moderate-carbohydrate, low-fat, low-glycemic index (GI) and low calorific products in appropriate portions will be encouraged. This diet will result in a relative increase in energy consumption from proteins, which also will promote satiety. Each patient will be provided with two booklets, one for food portion size exchange and tips for eating out, and another listing the low-GI food options and meal plans (GI <55). Furthermore, techniques for coping at-risk situations such as parties and festival celebrations will be taught. Recipes will also be provided to the patients to encourage healthy cooking. Adherence to dietary intervention will be assessed by calculating the percentage attendance to the intervention sessions and evaluating the dietary intakes and meal patterns using a weekly food record.

Besides, patients will be encouraged to see an exercise instructor at least once during the lifestyle modification programme. During the first exercise consultation (about 30 min), the exercise instructor will review the patient's medical history and exercise habits, and design a suitable exercise regime for the patient. The patients will first be instructed to do moderate intensity aerobic exercise for 30 min, 3 to 5 days a week and encouraged to increase daily physical activities.

During subsequent appointments, the exercise instructor will evaluate the patient's exercise progress on aerobic exercise and stretching during follow-ups. When the patients will be able to develop a routine exercise habit, they will be instructed to perform resistance training to increase their muscle endurance and strength for better aerobic performance and liver fat reduction (30). The intensity of exercise will be gradually increased to 30 minutes every day. The target will be a reduction of body mass index (BMI) towards 23 kg/m2.

Control group Patients in the control group will receive routine care at the medical clinic of the Prince of Wales Hospital, Hong Kong. At baseline, a clinician will explain the laboratory test results and the natural history of NAFLD to the patients. The patients will be encouraged to reduce carbohydrate and fat intake, and to exercise for at least 3 times per week, 30 minutes per session.

Follow up assessments in all groups The patients will attend the clinic at months 4 and 12 for metabolic assessment, and receive further advice from a clinician as appropriate. Before each visit, patients will be asked to fast overnight for at least 8 hours, then blood samples will be taken for liver biochemistry, glucose, insulin and lipids. Insulin resistance will be estimated using the homeostasis model assessment (HOMA-IR) calculated as fasting plasma glucose (mmol/L) x insulin (mIU/L) / 22.5 and quantitative insulin-sensitivity check index (QUICKI), calculated as 1/ [log fasting insulin (μU/mL) +log fasting glucose (mg/dL)]). Alanine aminotransferase (IU/L), fasting glucose (mmol/L), hemoglobin A1c (%), total cholesterol LDL, HDL(mmol/L) and triglycerides (mmol/L) will also be measured. Additionally, Weight, height will be measured during their clinical visit before each of their MRI scan and BMI will be calculated by weight (kg) / height^2 (m). Waist circumference will be measured at a level midway between the lower rib margin and iliac crest with the tape all around the body in the horizontal position. Physical activities will be recorded as the total duration of active exercise (min) per week.

Image Acquisition Subjects from all the groups will undergo MRI at baseline before their intervention and two follow-up scans at 4-months and 12-months intervals. All scanning will be performed using a Philips Achieva 3.0 Tesla MRI Scanner (Philips Medical System, Best, The Netherlands). Chemical-shift water-fat images will be acquired by the 3D spoiled multi-echo modified DIXON sequence with a 16-channel SENSE-XL-Torso array also from Philips Healthcare. Imaging parameters as follow: Repetition Time(TR) = 5.7-5.9 (ms), Echo time (TE)/echo spacing = 1.2-1.4 (ms) / 1.0-1.2 (ms), number of echoes = 6, flip angle = 3°, SENSE acceleration = 2, reconstructed slice thickness/number of slices = 3.0 mm / 50 to yield co-registered water, fat, fat-fraction and T2* image series. Non-breath-hold acquisition will be performed from the base of the skull to the base of the thoracic cavity for BAT measurement and breath-hold acquisition will be performed from the dome of the diaphragm to the pubic symphysis for abdominal SAT and VAT measurements.

T1 liver images will be acquired using 3D T1-fast-field echo (FFE) sequence, 2-echoes: TE1=1.8 msec, TE2=4.0 msec, TR=5.2 msec, flip angle=15, SENSE parallel imaging with acceleration factor 2.0 in phase-encoding direction.

In vivo quantification of liver fat will be performed using single voxel STEAM spectroscopy (TE=15 ms, TR=5000 ms, Number of signal avaregaes (NSA)=24, spectral width=2000 Hz, no water suppression). A 30×30×30-mm^3 (27 mL) voxel will be located on the right liver lobe to avoid major vessels according to the institutional protocol for hepatic fat measurement. Short TE and long TR will be selected to minimize T2 and T1 effects. Non-breath hold scan will be carried out and the acquisition time will be approximately 2 min.

Quantitative Measurement of Brown and Abdominal White Adipose Tissues Volume Brown adipose tissue (BAT) will be extracted from MR images using an in-house algorithm that has been validated and published in a recognized domain journal. This method utilizes the unique features of fat-fraction and T2* values in BAT to segment the tissue. Volume of BAT will be measured in mm^3 and be converted to mL.

Abdominal white adipose tissue will be separated into subcutaneous and visceral adipose tissues (SAT and VAT) using another in-house algorithm which has also been validated and published in a domain journal. Volume will be measured in mililitre (ml) and region of interest will be covered from the dome of diaphragm to the pubic symphysis.

Spectrum Analysis for Intrahepatic Triglycerides (IHTG). Magnetic resonance spectroscopy (MRS) data will be exported for offline time-domain analysis using the AMARES algorithm with Gaussian line shapes fitting in jMRUI software package. IHTG will be measured for relative fat signal integrals in terms of a percentage of the total signal amplitude. IHTG content is calculated as [signal Intensity of fat/(Signal Intensity of fat+Signal Intensity of water)] x 100. The definition of NAFLD will be based on liver fat content higher than the threshold of 5.5%.

Liver Inflammation and Fibrosis Liver inflammation and fibrosis (LIF) scores based on iron-corrected T1 (cT1) and T2* values will be calculated using LiverMultiScan™ (LMS, Perspectum Diagnostics, Oxford, UK). LIF scores range from 0-4 which 0 indicates the least severe and 4 as the most severe as show in figure 3. To validate the LIF scores, liver biopsy will be performed during the bariatric surgeries for assessment of degree of inflammation and fibrosis within the liver in association with NAFLD.

Statistical Analysis Within groups comparison will be measured using repeated measures ANOVA for results acquired from 3 different time points (baseline, Month 4 and Month 12). Variables with significant differences will be carried forward for pairwise comparison with bonferroni correction. Between groups comparison (life-style intervention and bariatric groups) will be measured in relative changes between baseline to Month 4 and Month 4 to Month12. Statistical analyses will be conducted using Statistical Package for the Social Sciences (SPSS) 25 (IBM, New York , USA). Significant level is selected at p < 0.05 (2-tailed).

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 25-30 kg/m2
* BMI ≥ 30 kg/m2 with Metabolic syndrome
* BMI ≥ 35 kg/m2 for morbid obesity

Exclusion Criteria:

* Other kind of hepatic diseases
* Under medications known to affect liver fat
* Waist circumference ≥ 150 cm
* Weight ≥ 250 kg
* MRI contraindications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Use of modified Dixon Magnetic Resonance Imaging method to measure the response of adipose tissue in different organs following life style modification program or Bariatric surgery | one year
  Abdominal subcutaneous fat in milliliters
Use of modified Dixon Magnetic Resonance Imaging method to measure the response of adipose tissue in different organs following life style modification program or Bariatric surgery 2 | one year
  Abdominal Visceral fat in milliliters
Use of modified Dixon Magnetic Resonance Imaging method to measure the response of adipose tissue in different organs following life style modification program or Bariatric surgery- 3 | one year
  Liver fat in percentage (%).
Use of modified Dixon Magnetic Resonance Imaging method to measure the response of adipose tissue in different organs following life style modification program or Bariatric surgery- 4 | one year
  pancreatic fat in percentage (%).
Use of modified Dixon Magnetic Resonance Imaging method to assess the relationship between Brown Adipose Tissue and Non Alcoholic Fatty Liver Disease | one year
  Brown fat in milliliters
Blood biochemistry for assessing β-cell function and insulin resistance (IR) | one year
  Homeostatic model assessment (HOMA) (Fasting glucose in nanomoles per liter (nmol/L) and insulin in (micro-units Per Litre).
Blood biochemistry- 1 | one year
  To measure Triglycerides in millimoles per litre (mmol/L)
Blood biochemistry- 2 | one year
  To measure high density lipoproteins in millimoles per litre (mmol/L)
Blood biochemistry- 3 | one year
  To measure Low-Density Lipoproteins in millimoles per litre (mmol/L)
Blood biochemistry- 4 | one year
  To measure ALT in International Units Per Litre (IU/L)
Blood biochemistry- 5 | one year
  To measure AST in International Units Per Litre (IU/L)
Blood biochemistry- 6 | one year
  To measure gamma-glutamyltransferase (GGT) in International Units Per Litre (IU/L)
Anthropomorphic measurements using measuring tape and weight scale | one year
  BMI in kg/m^2 (weight in kg and height in meters)
Anthropomorphic measurements using BP machine | one year
  Systolic and Diastolic Blood pressure in millimeters of mercury (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Winnie C Chu, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Prince of Wale Hospital, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szczepaniak LS, Nurenberg P, Leonard D, Browning JD, Reingold JS, Grundy S, Hobbs HH, Dobbins RL. Magnetic resonance spectroscopy to measure hepatic triglyceride content: prevalence of hepatic steatosis in the general population. Am J Physiol Endocrinol Metab. 2005 Feb;288(2):E462-8. doi: 10.1152/ajpendo.00064.2004. Epub 2004 Aug 31. PMID 15339742
- [Background] Wong VW, Wong GL, Yeung DK, Lau TK, Chan CK, Chim AM, Abrigo JM, Chan RS, Woo J, Tse YK, Chu WC, Chan HL. Incidence of non-alcoholic fatty liver disease in Hong Kong: a population study with paired proton-magnetic resonance spectroscopy. J Hepatol. 2015 Jan;62(1):182-9. doi: 10.1016/j.jhep.2014.08.041. Epub 2014 Sep 6. PMID 25195550
- [Background] Wong VW, Chu WC, Wong GL, Chan RS, Chim AM, Ong A, Yeung DK, Yiu KK, Chu SH, Woo J, Chan FK, Chan HL. Prevalence of non-alcoholic fatty liver disease and advanced fibrosis in Hong Kong Chinese: a population study using proton-magnetic resonance spectroscopy and transient elastography. Gut. 2012 Mar;61(3):409-15. doi: 10.1136/gutjnl-2011-300342. Epub 2011 Aug 16. PMID 21846782
- [Background] Bril F, Barb D, Portillo-Sanchez P, Biernacki D, Lomonaco R, Suman A, Weber MH, Budd JT, Lupi ME, Cusi K. Metabolic and histological implications of intrahepatic triglyceride content in nonalcoholic fatty liver disease. Hepatology. 2017 Apr;65(4):1132-1144. doi: 10.1002/hep.28985. Epub 2017 Feb 25. PMID 27981615
- [Background] Korenblat KM, Fabbrini E, Mohammed BS, Klein S. Liver, muscle, and adipose tissue insulin action is directly related to intrahepatic triglyceride content in obese subjects. Gastroenterology. 2008 May;134(5):1369-75. doi: 10.1053/j.gastro.2008.01.075. Epub 2008 Jan 30. PMID 18355813
- [Background] Fabbrini E, Magkos F, Mohammed BS, Pietka T, Abumrad NA, Patterson BW, Okunade A, Klein S. Intrahepatic fat, not visceral fat, is linked with metabolic complications of obesity. Proc Natl Acad Sci U S A. 2009 Sep 8;106(36):15430-5. doi: 10.1073/pnas.0904944106. Epub 2009 Aug 24. PMID 19706383
- [Background] Leong A, Porneala B, Dupuis J, Florez JC, Meigs JB. Type 2 Diabetes Genetic Predisposition, Obesity, and All-Cause Mortality Risk in the U.S.: A Multiethnic Analysis. Diabetes Care. 2016 Apr;39(4):539-46. doi: 10.2337/dc15-2080. Epub 2016 Feb 16. PMID 26884474
- [Background] Cypess AM, Kahn CR. Brown fat as a therapy for obesity and diabetes. Curr Opin Endocrinol Diabetes Obes. 2010 Apr;17(2):143-9. doi: 10.1097/MED.0b013e328337a81f. PMID 20160646
- [Background] Koksharova E, Ustyuzhanin D, Philippov Y, Mayorov A, Shestakova M, Shariya M, Ternovoy S, Dedov I. The Relationship Between Brown Adipose Tissue Content in Supraclavicular Fat Depots and Insulin Sensitivity in Patients with Type 2 Diabetes Mellitus and Prediabetes. Diabetes Technol Ther. 2017 Feb;19(2):96-102. doi: 10.1089/dia.2016.0360. PMID 28118051
- [Background] Donohoe CL, Doyle SL, Reynolds JV. Visceral adiposity, insulin resistance and cancer risk. Diabetol Metab Syndr. 2011 Jun 22;3:12. doi: 10.1186/1758-5996-3-12. PMID 21696633
- [Background] Cannon B, Nedergaard J. Brown adipose tissue: function and physiological significance. Physiol Rev. 2004 Jan;84(1):277-359. doi: 10.1152/physrev.00015.2003. PMID 14715917
- [Background] van Marken Lichtenbelt WD, Vanhommerig JW, Smulders NM, Drossaerts JM, Kemerink GJ, Bouvy ND, Schrauwen P, Teule GJ. Cold-activated brown adipose tissue in healthy men. N Engl J Med. 2009 Apr 9;360(15):1500-8. doi: 10.1056/NEJMoa0808718. PMID 19357405
- [Background] Cypess AM, Lehman S, Williams G, Tal I, Rodman D, Goldfine AB, Kuo FC, Palmer EL, Tseng YH, Doria A, Kolodny GM, Kahn CR. Identification and importance of brown adipose tissue in adult humans. N Engl J Med. 2009 Apr 9;360(15):1509-17. doi: 10.1056/NEJMoa0810780. PMID 19357406
- [Background] Wang Q, Zhang M, Xu M, Gu W, Xi Y, Qi L, Li B, Wang W. Brown adipose tissue activation is inversely related to central obesity and metabolic parameters in adult human. PLoS One. 2015 Apr 20;10(4):e0123795. doi: 10.1371/journal.pone.0123795. eCollection 2015. PMID 25894250
- [Background] Virtanen KA, Lidell ME, Orava J, Heglind M, Westergren R, Niemi T, Taittonen M, Laine J, Savisto NJ, Enerback S, Nuutila P. Functional brown adipose tissue in healthy adults. N Engl J Med. 2009 Apr 9;360(15):1518-25. doi: 10.1056/NEJMoa0808949. PMID 19357407
- [Background] Bartelt A, Heeren J. Adipose tissue browning and metabolic health. Nat Rev Endocrinol. 2014 Jan;10(1):24-36. doi: 10.1038/nrendo.2013.204. Epub 2013 Oct 22. PMID 24146030
- [Background] Purnak T, Ozaslan E. Brown adipose tissue: a novel marker for non-alcoholic fatty liver disease. Med Hypotheses. 2009 Nov;73(5):864. doi: 10.1016/j.mehy.2009.04.010. Epub 2009 May 17. No abstract available. PMID 19447565
- [Background] Yilmaz Y, Ones T, Purnak T, Ozguven S, Kurt R, Atug O, Turoglu HT, Imeryuz N. Association between the presence of brown adipose tissue and non-alcoholic fatty liver disease in adult humans. Aliment Pharmacol Ther. 2011 Aug;34(3):318-23. doi: 10.1111/j.1365-2036.2011.04723.x. Epub 2011 Jun 1. PMID 21631560
- [Background] Bartelt A, Bruns OT, Reimer R, Hohenberg H, Ittrich H, Peldschus K, Kaul MG, Tromsdorf UI, Weller H, Waurisch C, Eychmuller A, Gordts PL, Rinninger F, Bruegelmann K, Freund B, Nielsen P, Merkel M, Heeren J. Brown adipose tissue activity controls triglyceride clearance. Nat Med. 2011 Feb;17(2):200-5. doi: 10.1038/nm.2297. Epub 2011 Jan 23. PMID 21258337
- [Background] Ozguven S, Ones T, Yilmaz Y, Turoglu HT, Imeryuz N. The role of active brown adipose tissue in human metabolism. Eur J Nucl Med Mol Imaging. 2016 Feb;43(2):355-361. doi: 10.1007/s00259-015-3166-7. Epub 2015 Aug 19. PMID 26283505
- [Background] Scheja L, Heeren J. Metabolic interplay between white, beige, brown adipocytes and the liver. J Hepatol. 2016 May;64(5):1176-1186. doi: 10.1016/j.jhep.2016.01.025. Epub 2016 Jan 30. PMID 26829204
- [Background] Wei JL, Leung JC, Loong TC, Wong GL, Yeung DK, Chan RS, Chan HL, Chim AM, Woo J, Chu WC, Wong VW. Prevalence and Severity of Nonalcoholic Fatty Liver Disease in Non-Obese Patients: A Population Study Using Proton-Magnetic Resonance Spectroscopy. Am J Gastroenterol. 2015 Sep;110(9):1306-14; quiz 1315. doi: 10.1038/ajg.2015.235. Epub 2015 Jul 28. PMID 26215532
- [Background] Wong VW, Chan RS, Wong GL, Cheung BH, Chu WC, Yeung DK, Chim AM, Lai JW, Li LS, Sea MM, Chan FK, Sung JJ, Woo J, Chan HL. Community-based lifestyle modification programme for non-alcoholic fatty liver disease: a randomized controlled trial. J Hepatol. 2013 Sep;59(3):536-42. doi: 10.1016/j.jhep.2013.04.013. Epub 2013 Apr 23. PMID 23623998
- [Background] Wong VW, Wong GL, Chan RS, Shu SS, Cheung BH, Li LS, Chim AM, Chan CK, Leung JK, Chu WC, Woo J, Chan HL. Beneficial effects of lifestyle intervention in non-obese patients with non-alcoholic fatty liver disease. J Hepatol. 2018 Dec;69(6):1349-1356. doi: 10.1016/j.jhep.2018.08.011. Epub 2018 Aug 22. PMID 30142427
- [Background] Hui SCN, Wong SKH, Ai Q, Yeung DKW, Ng EKW, Chu WCW. Observed changes in brown, white, hepatic and pancreatic fat after bariatric surgery: Evaluation with MRI. Eur Radiol. 2019 Feb;29(2):849-856. doi: 10.1007/s00330-018-5611-z. Epub 2018 Jul 30. PMID 30062524
- [Background] Hui SCN, Ko JKL, Zhang T, Shi L, Yeung DKW, Wang D, Chan Q, Chu WCW. Quantification of brown and white adipose tissue based on Gaussian mixture model using water-fat and T2* MRI in adolescents. J Magn Reson Imaging. 2017 Sep;46(3):758-768. doi: 10.1002/jmri.25632. Epub 2017 Jan 16. PMID 28092409
- [Background] Hui SCN, Zhang T, Shi L, Wang D, Ip CB, Chu WCW. Automated segmentation of abdominal subcutaneous adipose tissue and visceral adipose tissue in obese adolescent in MRI. Magn Reson Imaging. 2018 Jan;45:97-104. doi: 10.1016/j.mri.2017.09.016. Epub 2017 Oct 7. PMID 29017799
- [Background] Wheeler ML, Franz M, Barrier P, Holler H, Cronmiller N, Delahanty LM. Macronutrient and energy database for the 1995 Exchange Lists for Meal Planning: a rationale for clinical practice decisions. J Am Diet Assoc. 1996 Nov;96(11):1167-71. doi: 10.1016/S0002-8223(96)00299-4. PMID 8906142
- [Background] Hallsworth K, Fattakhova G, Hollingsworth KG, Thoma C, Moore S, Taylor R, Day CP, Trenell MI. Resistance exercise reduces liver fat and its mediators in non-alcoholic fatty liver disease independent of weight loss. Gut. 2011 Sep;60(9):1278-83. doi: 10.1136/gut.2011.242073. Epub 2011 Jun 27. PMID 21708823